CLINICAL TRIAL: NCT07364461
Title: Diagnostic Accuracy of IgA Anti-transglutaminase Antibodies Measured by CLIA for Predicting Villous Atrophy in Coeliac Disease
Status: Completed | Type: Observational
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: P/23-168
Record Dates: First submitted 2026-01-13; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Coeliac Disease
Keywords: biopsy-free diagnosis; chemiluminescence immunoassays (CLIA); IgA anti-tissue transglutaminase 2 antibodies (TGA)
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CD patients
- Control

SUMMARY:
Celiac disease (CD) is an autoimmune disorder in which ingestion of gluten leads to immune-mediated damage of the small intestine. Diagnosis has traditionally required histological confirmation of duodenal villous atrophy.

Since 2012, European guidelines have allowed a biopsy-free diagnosis in paediatric patients with IgA anti-tissue transglutaminase 2 antibodies (TGA) levels greater than 10 times the upper limit of normal (>10 × ULN). In 2025, the diagnostic guidelines for adult CD included the possibility of biopsy-free diagnosis in patients younger than 45 years presenting TGA >10 × ULN, confirmed in a second serum sample. In both paediatric and adult guidelines, the supporting evidence was based almost exclusively on enzyme immunoassays (EIA) using chromogenic substrates such as ELISA or fluorogenic substrates such as FEIA.

In recent years, chemiluminescence immunoassays (CLIA) have largely replaced EIA in routine clinical practice. However, the optimal threshold for CD screening and for biopsy-free diagnosis using CLIA remains unclear, and the few available studies suggest values substantially higher than those established for EIA. Differences in analytical performance, wide variability in cut-off values, potential sex differences and limited real-world data raise concerns about the direct application of the >10 × ULN criterion to CLIA assays.

The primary aim of this study is to evaluate, in a community setting, the performance of CLIA-based TGA measurement to establish a threshold with high specificity and positive predictive value for duodenal villous atrophy (Marsh 2-3) suitable for biopsy-free CD diagnosis and to evaluate potential age and sex-related differences. The secondary aims are: 1) to determine the optimal cut-off for CD with duodenal atrophy screening; 2) to assess the accuracy of the manufacturer recommended cut-off.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone duodenal biopsy and a complete CD diagnostic work-up
* Eating a gluten-containing diet

Exclusion Criteria:

* Having an unsuitable or non-performed duodenal biopsy
* Incomplete clinical data
* Inconclusive diagnostic findings
* Previous diagnosis of CD with duodenal biopsy performed during gluten-free diet (GFD)
* IgA deficiency

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had TGA measured by CLIA within the healthcare area served by the Catlab Clinical Analysis Laboratory, covering a population of 717.181 inhabitants as of 1 January 2024 (IDESCAT). This area includes primary care centres and three community hospitals: University Hospital Mútua Terrassa, University Hospital Consorci Sanitari de Terrassa and Consorci Corporació Sanitària Parc Taulí.
Sampling Method: Probability Sample
Enrollment: 765 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Optimal cut-off value of TGA levels measured by CLIA for biopsy-free CD diagnosis | Baseline
  The optimal TGA cut-off value for CD diagnosis with duodenal atrophy will be determined using the cost function minimization method to achieve positive predictive values and specificities of over 95%

CONTACTS AND LOCATIONS:
Locations (1):
- CatLab AIE, Viladecavalls, Barcelona, Spain